CLINICAL TRIAL: NCT01768962
Title: A Phase 1 Crossover Trial Evaluating the Pharmacokinetics of Tenofovir Reduced-Glycerin 1% Gel in the Rectal and Vaginal Compartments in Women
Brief Title: Tenofovir Levels Following Local Application of Tenofovir Reduced-Glycerin 1% Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MTN-014; 5UM1AI068633 (NIH); 11885 (Other Grant/Funding Number: DAIDS Protocol Number)
Record Dates: First submitted 2012-11-20; First posted 2013-01-16 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: HIV Prevention
Keywords: Microbicides; Tenofovir; Reduced-glycerin; Vaginal use; Rectal use; Pharmacokinetics
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence A (Active Comparator): 2 weeks, 6 week washout, 2 weeks
  Interventions: Drug: Once Daily Application of TFV RG 1% Gel - Vaginal; Drug: Once Daily Application of TFV RG 1% gel - Rectal
- Sequence B (Active Comparator): 2 weeks, 6 week washout, 2 weeks
  Interventions: Drug: Once Daily Application of TFV RG 1% gel - Rectal; Drug: Once Daily Application of TFV RG 1% Gel - Vaginal

INTERVENTIONS:
Drug: Once Daily Application of TFV RG 1% Gel - Vaginal — Vaginal application
  Arms: Sequence A
Drug: Once Daily Application of TFV RG 1% gel - Rectal — Rectal application
  Arms: Sequence A
Drug: Once Daily Application of TFV RG 1% gel - Rectal — Rectal application
  Arms: Sequence B
Drug: Once Daily Application of TFV RG 1% Gel - Vaginal — Vaginal application
  Arms: Sequence B

SUMMARY:
To compare local and systemic pharmacokinetics of tenofovir reduced-glycerin (TFV RG) 1% gel after 2 weeks of daily rectal use and after 2 weeks of daily vaginal use

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 through 45 years (inclusive) at Screening
2. Able and willing to provide written informed consent
3. Able and willing to comply with all study procedure requirements, including, clinical and laboratory assessments, vaginal and rectal examinations, urine and blood testing, as well as attendance at all scheduled study visits
4. In general good health at Screening and Enrollment as determined by the Investigator of Record (IoR)/ or designee
5. Negative pregnancy test at Screening and Enrollment
6. HIV-negative at Screening and Enrollment
7. Able and willing to provide adequate locator information
8. Willingness to use study-provided male condoms for the duration of study participation for penetrative intercourse
9. Per participant report at Screening, regular menstrual cycles with at least 21 days between menses (does not apply to participants who report using a progestin-only method of contraception at screening, e.g., Depo-Provera, progesterone-containing IUDs or extended use of oral contraceptives)
10. Per participant report at Enrollment, using an effective method of contraception and intending to use an effective method for the duration of study participation; effective methods include:

    * Hormonal methods, excluding vaginal rings
    * Intrauterine device (IUD) inserted at least 42 days prior to Enrollment (but not past the maximum length of recommended usage according to package instructions)
    * Sterilization of participant or partner at least 42 days prior to Enrollment
    * Self-identifies as a woman who has sex with women exclusively
    * Sexually abstinent for the at least 90 days prior to enrollment and the intention to remain sexually abstinent for the duration of study participation
11. Per participant report at Screening, states a willingness to refrain from inserting any non-study vaginal or rectal products or objects into the vagina or rectum, including but not limited to, spermicides, female condoms, diaphragms, contraceptive vaginal rings, vaginal medications, menstrual cups, cervical caps (or any other vaginal barrier method), vaginal/rectal douches, enemas, non-study approved lubricants, sex toys (vibrators, dildos, etc.), and tampons for the duration of the study product use periods and for 24 hours prior to each scheduled study clinic visit.
12. Pap result consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009) or satisfactory evaluation of non-Grade 0 Pap result with no treatment required per clinical judgment of IoR or designee in the 12 calendar months prior to the Enrollment Visit
13. At Screening, participant agrees not to take part in other research studies involving drugs, medical devices, or vaginal/rectal products for the duration of study participation (including the time between the Screening and Enrollment visits)

    Participants in the biopsy subset must also meet the following criteria at Screening to be eligible for inclusion:
14. Willing to abstain from inserting anything into the vagina or rectum for 72 hours prior to and following the collection of these samples, including vaginal and rectal intercourse
15. Willing to restrict the use of non-steroidal anti-inflammatory drugs (NSAIDs), aspirin and/or other drugs that are associated with the increased likelihood of bleeding following mucosal biopsy collection for 72 hours prior to and following the collection biopsies

Exclusion Criteria:

1. Participant report of any of the following:

   1. Known adverse reaction to the study product (ever)
   2. Known adverse reaction to latex (ever)
   3. Current male sex partner with known history of adverse reaction to latex (ever)
   4. History of serum HBsAg positivity (ever)
   5. Non-therapeutic injection drug use in the 12 calendar months prior to Enrollment
   6. Sexually transmitted infections (STI) or reproductive tract infection (RTI) requiring treatment in the 6 calendar months prior to Enrollment
   7. Post-exposure prophylaxis (PEP) for possible HIV-1 infection within the 6 calendar months prior to Enrollment
   8. Last pregnancy outcome within 90 days or less prior to Enrollment
   9. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage) within the 42 days prior to Enrollment Note: This does not include biopsy for the evaluation of an abnormal pap result or endometrial biopsy that occurred more than 7 days prior to Enrollment, provided that all other inclusion/exclusion criteria are met.
   10. Participation in any other research study involving drugs, medical devices or vaginal products 42 days or less prior to Enrollment
   11. Anticipated IUD replacement within the next 3 months or an IUD inserted 42 days or less prior to Enrollment
   12. Participant report at Screening and/or Enrollment intention of becoming pregnant in the next 3 months
   13. Currently breastfeeding at the time of Screening and/or Enrollment
   14. History of bleeding problems (Participants in the biopsy subset only)
2. Laboratory abnormalities at Screening greater than or equal to a Grade 2*:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT)
   2. Hemoglobin
   3. Platelet count
   4. Serum creatinine Otherwise eligible participants with an exclusionary test result(s) listed above may be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within the 42 days of providing informed consent, the participant may be enrolled.
3. Urinary tract infection (UTI) at Screening and/or Enrollment Note: Otherwise eligible participants diagnosed with UTI during Screening will be offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 42 days of obtaining informed consent, the participant may be enrolled.
4. Pelvic inflammatory disease or an STI or RTI requiring treatment per current World Health Organization (WHO) guidelines at Screening and/or Enrollment
5. Clinically apparent Grade 2 or higher pelvic** and/or rectal*** examination finding (observed by study staff) at Screening and/or Enrollment Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.

   Note: Otherwise eligible participants with exclusionary pelvic and/or rectal examination findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved. If improvement to a non-exclusionary grade or resolution is documented within 42 days of providing informed consent, the participant may be enrolled.
6. Any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

   * per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009) ** per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009), Addendum 1 Female Genital Grading Table for Use in Microbicide Studies *** per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009), Addendum 3 Rectal Grading Table for Use in Microbicide Studies (Clarification dated May 2012).

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Drug concentrations | 10 weeks
  To compare local and systemic pharmacokinetics of tenofovir reduced-glycerin 1% gel after 2 weeks of daily rectal use and after 2 weeks of daily vaginal use

SECONDARY OUTCOMES:
Number of adverse events Grade 2 or higher | 10 weeks
  To assess the safety of tenofovir reduced-glycerin 1% gel after 2 weeks of daily rectal use and after 2 weeks of daily vaginal use

OTHER OUTCOMES:
Inhibition of HIV by study drug in rectal and genital fluids | 10 weeks
  Correlate drug levels in rectal and genital fluids with drug potency
Microflora biomarkers and gene expression from the vaginal and rectal environments | 10 weeks
  Determine changes in microflora biomarkers and gene expression from the vaginal and rectal environments after 2 weeks of daily rectal versus 2 weeks of daily vaginal use of tenofovir reduced-glycerin 1% gel at sites with capacity

CONTACTS AND LOCATIONS:
Overall Officials: Gonasagrie Nair, MBChB, Study Chair — Centre for the AIDS Programme of Research in South Africa (CAPRISA) - eThekwini CRS; Jessica Justman, MD, Principal Investigator — Columbia University
Locations (1):
- Center for Infectious Disease Epidemiologic Research, Mailman School of Public Health, Columbia University, New York, New York, United States

REFERENCES:
- [Background] Justman JE, Nair GL, Hendrix CW, Piper JM, Marzinke MA, Dai JY, Pan Z, Galaska B, Levy L, Schwartz JL, Balar B, Kunjara Na Ayudhya RP, Mushamiri I, McGowan I, Dezzutti CS; MTN-014 Study Team. Pharmacokinetics and Pharmacodynamics of Tenofovir Reduced-Glycerin 1% Gel in the Rectal and Vaginal Compartments in Women: A Cross-Compartmental Study With Directly Observed Dosing. J Acquir Immune Defic Syndr. 2018 Jun 1;78(2):175-182. doi: 10.1097/QAI.0000000000001655. PMID 29767639
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29767639